CLINICAL TRIAL: NCT05459714
Title: A Prospective Study to Evaluate the Feasibility and Safety of Magnetically Controlled Capsule Endoscope System in Stomach Examination of Moderately and Severely Obese Patients
Brief Title: Magnetically Controlled Capsule Endoscope System in Stomach Examination of Moderately and Severely Obese Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Changhai Hospital (Other)
Collaborators: Shanghai 6th People's Hospital (Other); Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other)
Responsible Party: Principal Investigator, Zhuan Liao, Professor, Changhai Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MCE for obese patients
Record Dates: First submitted 2022-07-11; First posted 2022-07-15 (Actual); Last update posted 2022-07-15 (Actual); Status verified 2022-07

CONDITIONS: Obesity
Keywords: obesity; capsule endoscopy
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MCE for obese patients (Experimental): After a standardized gastrointestinal preparation, the patient will undergo MCE examination. After completing the MCE procedure, the patient is evaluated for examination comfort and can then leave the hospital on his or her own and watch for capsule excretion.
  Interventions: Device: MCE for obese patients

INTERVENTIONS:
Device: MCE for obese patients — Sequence of stomach examination: The stomach examination is performed sequentially according to the order of fundus, cardia, gastric body, angulus, antrum, and pylorus, which should ensure the integrity of the observation of each part of the stomach and achieve the purpose of comprehensive observation by means of different observation distances such as distant view and close view, and different observation angles such as front and side.

SUMMARY:
This study is a prospective, multicenter clinical trial. The study is planned to be conducted at a qualified clinical trial center, and 30 subjects are planned to be enrolled to evaluate the feasibility and safety of magnetically controlled capsule endoscopy (MCE) system in the examination of gastric disorders in patients with moderate to severe obesity (BMI ≥ 35 kg/m2).

DETAILED DESCRIPTION:
Metabolic surgery, as one of the most important treatments for obesity, has been widely used worldwide. Esophagogastroduodenoscopy (EGD) is mostly used in the perioperative preoperative application of metabolic surgery to improve or exclude preoperative diagnosis, including gastrointestinal tumors, various types of upper GI mucosal lesions, esophagitis, esophageal hiatal hernia, gastrointestinal interstitial tumors, etc. However, EGD is an invasive examination and can cause discomfort without anesthesia, resulting in low patient compliance. In 2013, ANKON took the lead in developing the world's first capsule endoscope system that utilizes precise multi-dimensional rotational movement of a robotic arm and adaptive matching to achieve precise magnetic control, which is convenient for observing specific lesions from an appropriate angle and has been shown to have high diagnostic accuracy for gastric diseases (highly consistent with EGD, with sensitivity and specificity of 90.4% and 95.7%, respectively, and accuracy of 93.4%). It has been clinically proven that MCE is safe and effective in the upper gastrointestinal tract, but there is a lack of clinical systematic studies on its application to moderately and severely obese people.In summary, this exploratory study is designed to preliminarily verify the clinical feasibility and safety of MCE for upper gastrointestinal examination in moderately obese people (BMI ≥ 35 kg/m2).

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of obesity: BMI ≥ 35kg/m2;
2. Be scheduled to undergo gastric examination;
3. Be able to provide informed consent.

Exclusion Criteria:

1. With swallowing obstruction or disorders; 2. With known or suspected gastrointestinal obstruction, stenosis and fistula; 3. Have no conditions for surgery or refuse to undergo any abdominal surgery; 4. Be allergic to or have other known contraindication or intolerance to the drug used in the study; 5. With pacemakers or other electronic devices such as electronic cochlear implants, implanted magnetic metal drug infusion pumps, neurostimulators, and magnetic metal foreign bodies; 6. Women during pregnancy; 7. Currently enrolled in another clinical trial of a drug or device; 8. Other conditions determined by the investigator to be inappropriate for enrollment.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-10-15 (Estimated); Primary Completion 2023-05-01 (Estimated); Study Completion 2023-05-01 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Complete Observation | 2 weeks
  The number of participants with complete observation. Complete observation of the mucosa means over 90% of the mucosa observed in gastric cardia, fundus, body, angulus, antrum and pylorus.

SECONDARY OUTCOMES:
Gastric Examination Time | 2 weeks
  Gastric examination time was defined as the time taken for the endoscopist to complete the gastric examination to his or her satisfaction
The Total Number of Patients Who Who Had a Diagnosis of Positive Findings | 2 weeks
  It was calculated using the following formula: number of patients with positive findings divided by the total number of patients that underwent examination.
Evaluation of patient satisfaction through questionaires | 2 weeks
  The investigators use a satisfaction questionnaire to evaluate the satisfaction of each patient, including ease of capsule swallowing, discomfort during the examination, discomfort after the examination and comfort level of MCE examination.

CONTACTS AND LOCATIONS:
Overall Officials: Pin Zhang, Principal Investigator — Shanghai 6th People's Hospital; Kai Yin, Principal Investigator — Changhai Hospital; Bin Wang, Principal Investigator — Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University
Locations (3):
- China (3):
  - Changhai Hospital, Shanghai
  - Shanghai Ninth People's Hospital, Shanghai
  - Shanghai Sixth People's Hospital, Shanghai

IPD SHARING:
Plan to Share IPD: Yes
After finishing this study, the investigators will make the data available to other researchers:
  including study protocol, statistical analysis plan (SAP), informed consent form (ICF), clinical study report (CSR)
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 3 years
Access Criteria: The website of the journal where the results published, and ClinicalTrials.gov web site.

REFERENCES:
- [Background] GBD 2015 Obesity Collaborators; Afshin A, Forouzanfar MH, Reitsma MB, Sur P, Estep K, Lee A, Marczak L, Mokdad AH, Moradi-Lakeh M, Naghavi M, Salama JS, Vos T, Abate KH, Abbafati C, Ahmed MB, Al-Aly Z, Alkerwi A, Al-Raddadi R, Amare AT, Amberbir A, Amegah AK, Amini E, Amrock SM, Anjana RM, Arnlov J, Asayesh H, Banerjee A, Barac A, Baye E, Bennett DA, Beyene AS, Biadgilign S, Biryukov S, Bjertness E, Boneya DJ, Campos-Nonato I, Carrero JJ, Cecilio P, Cercy K, Ciobanu LG, Cornaby L, Damtew SA, Dandona L, Dandona R, Dharmaratne SD, Duncan BB, Eshrati B, Esteghamati A, Feigin VL, Fernandes JC, Furst T, Gebrehiwot TT, Gold A, Gona PN, Goto A, Habtewold TD, Hadush KT, Hafezi-Nejad N, Hay SI, Horino M, Islami F, Kamal R, Kasaeian A, Katikireddi SV, Kengne AP, Kesavachandran CN, Khader YS, Khang YH, Khubchandani J, Kim D, Kim YJ, Kinfu Y, Kosen S, Ku T, Defo BK, Kumar GA, Larson HJ, Leinsalu M, Liang X, Lim SS, Liu P, Lopez AD, Lozano R, Majeed A, Malekzadeh R, Malta DC, Mazidi M, McAlinden C, McGarvey ST, Mengistu DT, Mensah GA, Mensink GBM, Mezgebe HB, Mirrakhimov EM, Mueller UO, Noubiap JJ, Obermeyer CM, Ogbo FA, Owolabi MO, Patton GC, Pourmalek F, Qorbani M, Rafay A, Rai RK, Ranabhat CL, Reinig N, Safiri S, Salomon JA, Sanabria JR, Santos IS, Sartorius B, Sawhney M, Schmidhuber J, Schutte AE, Schmidt MI, Sepanlou SG, Shamsizadeh M, Sheikhbahaei S, Shin MJ, Shiri R, Shiue I, Roba HS, Silva DAS, Silverberg JI, Singh JA, Stranges S, Swaminathan S, Tabares-Seisdedos R, Tadese F, Tedla BA, Tegegne BS, Terkawi AS, Thakur JS, Tonelli M, Topor-Madry R, Tyrovolas S, Ukwaja KN, Uthman OA, Vaezghasemi M, Vasankari T, Vlassov VV, Vollset SE, Weiderpass E, Werdecker A, Wesana J, Westerman R, Yano Y, Yonemoto N, Yonga G, Zaidi Z, Zenebe ZM, Zipkin B, Murray CJL. Health Effects of Overweight and Obesity in 195 Countries over 25 Years. N Engl J Med. 2017 Jul 6;377(1):13-27. doi: 10.1056/NEJMoa1614362. Epub 2017 Jun 12. PMID 28604169
- [Background] Praveenraj P, Gomes RM, Kumar S, Senthilnathan P, Parathasarathi R, Rajapandian S, Palanivelu C. Diagnostic Yield and Clinical Implications of Preoperative Upper Gastrointestinal Endoscopy in Morbidly Obese Patients Undergoing Bariatric Surgery. J Laparoendosc Adv Surg Tech A. 2015 Jun;25(6):465-9. doi: 10.1089/lap.2015.0041. Epub 2015 May 5. PMID 25942627
- [Background] Liao Z, Duan XD, Xin L, Bo LM, Wang XH, Xiao GH, Hu LH, Zhuang SL, Li ZS. Feasibility and safety of magnetic-controlled capsule endoscopy system in examination of human stomach: a pilot study in healthy volunteers. J Interv Gastroenterol. 2012 Oct-Dec;2(4):155-160. doi: 10.4161/jig.23751. Epub 2012 Oct 1. PMID 23687601
- [Background] Liao Z, Hou X, Lin-Hu EQ, Sheng JQ, Ge ZZ, Jiang B, Hou XH, Liu JY, Li Z, Huang QY, Zhao XJ, Li N, Gao YJ, Zhang Y, Zhou JQ, Wang XY, Liu J, Xie XP, Yang CM, Liu HL, Sun XT, Zou WB, Li ZS. Accuracy of Magnetically Controlled Capsule Endoscopy, Compared With Conventional Gastroscopy, in Detection of Gastric Diseases. Clin Gastroenterol Hepatol. 2016 Sep;14(9):1266-1273.e1. doi: 10.1016/j.cgh.2016.05.013. Epub 2016 May 20. PMID 27211503
- [Background] Jiang X, Qian YY, Liu X, Pan J, Zou WB, Zhou W, Luo YY, Chen YZ, Li ZS, Liao Z. Impact of magnetic steering on gastric transit time of a capsule endoscopy (with video). Gastrointest Endosc. 2018 Oct;88(4):746-754. doi: 10.1016/j.gie.2018.06.031. Epub 2018 Jul 11. PMID 30005825